CLINICAL TRIAL: NCT02498119
Title: The Role of Arachidonic Acid Metabolites, in the Lipid Droplets of Macrophages From Patients With Metabolic Syndrome
Brief Title: The Role of Arachidonic Acid Metabolites, From Patients With Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Gracie Ong @ Gracie Ong Siok Yan, Senior Consultant, University of Malaya
Other Study IDs: RG291-14AFR
Record Dates: First submitted 2015-05-14; First posted 2015-07-15 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 DM; lipid bodies
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Whole blood is collected and blood component separated for the future use. Whole blood, red blood cells, plasma and buffy coat are was separated and kept in -80 degree Celsius.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Patient sample within the normal range of blood results.
- Abnormal: Patient sample from freshly diagnosed Type 2 Diabetes Mellitus.

SUMMARY:
The purpose of this study is to determine whether an increase in lipid bodies in leukocytes will lead to an increase in eicosanoid production. The 2nd purpose is to determine if there is a significant correlation between lipid body formation and enhanced generation of both Lipoxygenase (LO) and COX derived eicosanoids. The 3rd purpose is, if lipid bodies are involved in arachidonic acid (AA) metabolism, then AA present in these lipid rich structure must be released by phospholipases and the free Arachidonic Acid (AA) must have access to the eicosanoid forming enzyme. The fourth objective is to determine the compartmentalisation of cPLA2 and MAP kinases including ERK1, ERK2, p85 and p38 are involved in AA liberation within lipid bodies.

DETAILED DESCRIPTION:
Metabolic syndrome is a cluster of biochemical and physiological abnormalities associated with the development of cardiovascular disease and type 2 diabetes mellitus. The current study focused on type 2 Diabetes Mellitus(T2DM). T2DM is a chronic disease in which people have problems regulating their blood sugar. This disorder consists of an array of dysfunctions characterized by hyperglycemia and resulting from the combination of resistance of insulin action, inadequate insulin secretion and excessive or inappropriate glucagon secretion. Insulin resistance results from a complex interplay between nutrient overload, systemic fatty acid excess, inflammation of the adipose tissue, endoplasmic reticulum and oxidative stress.

At the molecular lever, inflammatory cytokines, fatty acid derivatives such as ceramides, diacylglycerols and reactive oxygen species (ROS), activate several serine/threonine kinases, that have emerged as important negative regulators of insulin signaling. Because of their ability to directly oxidize DNA, protein and lipid damage, ROS are believed to play a key role in the metabolic syndrome and the possible development of T2DM. It is possible that ROS and oxidative stress, induced by elevations in glucose and possibly free fatty acid levels play a key role in causing insulin resistance, and beta cell dysfunction by their ability to activate stress sensitive signaling pathways.

Lipids as signaling intermediates encompass a vast range of molecules with distinct function. The characteristics includes, lipid bodies(LB) are sites for the production of inflammatory mediators and LB within inflammatory cells contain arachidonyl lipids which serve as precursors for eicosanoids. In addition, formation of LB within inflammatory macrophages was positively correlated with augmented increase in prostaglandin E2 (PGE2) in changes. LB also could function as a draining compartment to rapidly uptake and re-acetylate free arachidonic acid with the potentially detrimental outcomes for the host cell.

Macrophage from cells with lipid bodies involves complex and multi step mechanisms that depend on different signaling pathways regulating lipid influx, metabolism storage and mobilization. In view of these clues the investigators have reason to believe that organic anion transporters might be resident or upon stimulation trans located to lipid bodies in order to export the newly synthesized lipid mediators into the cytoplasmic space. Once outside the lipid bodies the eicosanoids can exert intracrine functions or be exported to plasma membrane resident transporters to the extracellular space. Free fatty acids have adverse effects on the mitochondrial function including uncoupling of oxidative phosphorylation and the generation of ROS. Beta cell lipotoxicity has an amplifying effect only if mediated by concurrent hyperglycemia. The association of obesity, fatty acids and oxidative stress with insulin action clearly merits further attention with particular focus on the molecular mechanism.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 to ≤ 60
* Patient diagnosed with Type 2 Diabetes Mellitus within 1 year

Exclusion Criteria:

* Patients < 18 years
* Patients with uncontrolled diabetes, heart failure and sepsis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study subjects are recruited from Primary Care Clinic of University Malaya Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Composite measure of patient physical observations to include weight, height and BMI | six months only (1 time only)

SECONDARY OUTCOMES:
Reduction of pro - inflammatory cytokines | one year
The effect of eicosanoids in diabetic complication | One year
The effect of LTB4 and LTC4 of eicosanoids | One year

CONTACTS AND LOCATIONS:
Overall Officials: Gracie Ong Siok Yan, Principal Investigator — Senior Consultant
Locations (1):
- University Malaya Medical Center (UMMC), Petaling Jaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Melo RC, D'Avila H, Wan HC, Bozza PT, Dvorak AM, Weller PF. Lipid bodies in inflammatory cells: structure, function, and current imaging techniques. J Histochem Cytochem. 2011 May;59(5):540-56. doi: 10.1369/0022155411404073. Epub 2011 Mar 23. PMID 21430261
- [Background] Melo RC, Paganoti GF, Dvorak AM, Weller PF. The internal architecture of leukocyte lipid body organelles captured by three-dimensional electron microscopy tomography. PLoS One. 2013;8(3):e59578. doi: 10.1371/journal.pone.0059578. Epub 2013 Mar 26. PMID 23555714
- [Background] Tauchi-Sato K, Ozeki S, Houjou T, Taguchi R, Fujimoto T. The surface of lipid droplets is a phospholipid monolayer with a unique Fatty Acid composition. J Biol Chem. 2002 Nov 15;277(46):44507-12. doi: 10.1074/jbc.M207712200. Epub 2002 Sep 6. PMID 12221100
- [Background] Dichlberger A, Schlager S, Lappalainen J, Kakela R, Hattula K, Butcher SJ, Schneider WJ, Kovanen PT. Lipid body formation during maturation of human mast cells. J Lipid Res. 2011 Dec;52(12):2198-2208. doi: 10.1194/jlr.M019737. Epub 2011 Oct 4. PMID 21971714
- [Background] Krahmer N, Farese RV Jr, Walther TC. Balancing the fat: lipid droplets and human disease. EMBO Mol Med. 2013 Jul;5(7):973-83. doi: 10.1002/emmm.201100671. Epub 2013 Jun 6. PMID 23740690
- [Background] Hapala I, Marza E, Ferreira T. Is fat so bad? Modulation of endoplasmic reticulum stress by lipid droplet formation. Biol Cell. 2011 Jun;103(6):271-85. doi: 10.1042/BC20100144. PMID 21729000
- [Background] Beller M, Thiel K, Thul PJ, Jackle H. Lipid droplets: a dynamic organelle moves into focus. FEBS Lett. 2010 Jun 3;584(11):2176-82. doi: 10.1016/j.febslet.2010.03.022. Epub 2010 Mar 18. PMID 20303960
- [Background] Brasaemle DL. Thematic review series: adipocyte biology. The perilipin family of structural lipid droplet proteins: stabilization of lipid droplets and control of lipolysis. J Lipid Res. 2007 Dec;48(12):2547-59. doi: 10.1194/jlr.R700014-JLR200. Epub 2007 Sep 18. PMID 17878492
- [Background] Goodman JM. The gregarious lipid droplet. J Biol Chem. 2008 Oct 17;283(42):28005-9. doi: 10.1074/jbc.R800042200. Epub 2008 Jul 8. No abstract available. PMID 18611863
- [Background] Blaner WS, O'Byrne SM, Wongsiriroj N, Kluwe J, D'Ambrosio DM, Jiang H, Schwabe RF, Hillman EM, Piantedosi R, Libien J. Hepatic stellate cell lipid droplets: a specialized lipid droplet for retinoid storage. Biochim Biophys Acta. 2009 Jun;1791(6):467-73. doi: 10.1016/j.bbalip.2008.11.001. Epub 2008 Nov 24. PMID 19071229
- [Background] Dvorak AM, Dvorak HF, Peters SP, Shulman ES, MacGlashan DW Jr, Pyne K, Harvey VS, Galli SJ, Lichtenstein LM. Lipid bodies: cytoplasmic organelles important to arachidonate metabolism in macrophages and mast cells. J Immunol. 1983 Dec;131(6):2965-76. PMID 6315820
- [Background] Dvorak AM, Hammel I, Schulman ES, Peters SP, MacGlashan DW Jr, Schleimer RP, Newball HH, Pyne K, Dvorak HF, Lichtenstein LM, et al. Differences in the behavior of cytoplasmic granules and lipid bodies during human lung mast cell degranulation. J Cell Biol. 1984 Nov;99(5):1678-87. doi: 10.1083/jcb.99.5.1678. PMID 6436254
- [Background] Triggiani M, Oriente A, Marone G. Differential roles for triglyceride and phospholipid pools of arachidonic acid in human lung macrophages. J Immunol. 1994 Feb 1;152(3):1394-403. PMID 8301140
- [Background] Yu W, Bozza PT, Tzizik DM, Gray JP, Cassara J, Dvorak AM, Weller PF. Co-compartmentalization of MAP kinases and cytosolic phospholipase A2 at cytoplasmic arachidonate-rich lipid bodies. Am J Pathol. 1998 Mar;152(3):759-69. PMID 9502418
- [Background] Triggiani M, Oriente A, Seeds MC, Bass DA, Marone G, Chilton FH. Migration of human inflammatory cells into the lung results in the remodeling of arachidonic acid into a triglyceride pool. J Exp Med. 1995 Nov 1;182(5):1181-90. doi: 10.1084/jem.182.5.1181. PMID 7595189
- [Background] Silva AR, Pacheco P, Vieira-de-Abreu A, Maya-Monteiro CM, D'Alegria B, Magalhaes KG, de Assis EF, Bandeira-Melo C, Castro-Faria-Neto HC, Bozza PT. Lipid bodies in oxidized LDL-induced foam cells are leukotriene-synthesizing organelles: a MCP-1/CCL2 regulated phenomenon. Biochim Biophys Acta. 2009 Nov;1791(11):1066-75. doi: 10.1016/j.bbalip.2009.06.004. Epub 2009 Jun 30. PMID 19573621
- [Background] Bozza PT, Bakker-Abreu I, Navarro-Xavier RA, Bandeira-Melo C. Lipid body function in eicosanoid synthesis: an update. Prostaglandins Leukot Essent Fatty Acids. 2011 Nov;85(5):205-13. doi: 10.1016/j.plefa.2011.04.020. Epub 2011 May 12. PMID 21565480
- See also: The internal architecture of leukocyte lipid body organelles captured by three-dimensional electron microscopy tomography — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0059578
- See also: Lipid body formation during maturation of human mast cells — http://www.jlr.org/content/52/12/2198.long
- See also: Balancing the fat: lipid droplets and human disease — http://www.ncbi.nlm.nih.gov/pubmed/23740690
- See also: Is fat so bad? Modulation of endoplasmic reticulum stress by lipid droplet formation — http://www.ncbi.nlm.nih.gov/pubmed/21729000
- See also: a dynamic organelle moves into focus — http://www.ncbi.nlm.nih.gov/pubmed/20303960
- See also: The perilipin family of structural lipid droplet proteins: stabilization of lipid droplets and control of lipolysis — http://www.ncbi.nlm.nih.gov/pubmed/17878492
- See also: Hepatic stellate cell lipid droplets: a specialized lipid droplet for retinoid storage — http://www.ncbi.nlm.nih.gov/pubmed/19071229
- See also: Lipid bodies: cytoplasmic organelles important to arachidonate metabolism in macrophages and mast cells — http://www.ncbi.nlm.nih.gov/pubmed/6315820
- See also: Differences in the behavior of cytoplasmic granules and lipid bodies during human lung mast cell degranulation — http://www.ncbi.nlm.nih.gov/pubmed/6436254
- See also: Differential roles for triglyceride and phospholipid pools of arachidonic acid in human lung macrophages — http://www.ncbi.nlm.nih.gov/pubmed/8301140
- See also: Co-compartmentalization of MAP kinases and cytosolic phospholipase A2 at cytoplasmic arachidonate-rich lipid bodies — http://www.ncbi.nlm.nih.gov/pubmed/9502418
- See also: Migration of human inflammatory cells into the lung results in the remodeling of arachidonic acid into a triglyceride pool — http://www.ncbi.nlm.nih.gov/pubmed/7595189
- See also: Lipid bodies in oxidized LDL-induced foam cells are leukotriene-synthesizing organelles: a monocyte chemotactic protein 1/ chemokine ligand 2 (MCP-1/CCL2) regulated phenomenon — http://www.ncbi.nlm.nih.gov/pubmed/19573621
- See also: Lipid body function in eicosanoids synthesis : An update — http://www.ncbi.nlm.nih.gov/pubmed/21565480